CLINICAL TRIAL: NCT04236635
Title: A Phase 2B, Open-Label Study to Explore Tissue Histopathology Following Subcutaneous Injection of Collagenase Clostridium Histolyticum Using An Abdominoplasty Model
Brief Title: Histopathology Following CCH Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EN3835-213
Record Dates: First submitted 2020-01-02; First posted 2020-01-22 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Characteristics of Subcutaneous Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: CCH Single Injection Technique (Experimental): Participants were administered 0.07 milligrams (mg) CCH subcutaneously using a single injection technique.
  Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -43 and -22. Area 2 was administered CCH on Day -14.
  Interventions: Drug: Collagenase Clostridium Histolyticum Single Injection Technique
- Group 2: CCH Single Injection Technique (Experimental): Participants were administered 0.07 mg CCH subcutaneously using a single injection technique. Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -24 and -3. Area 2 was administered CCH on Day -3.
  Interventions: Drug: Collagenase Clostridium Histolyticum Single Injection Technique
- Group 3: CCH Single Injection Technique (Experimental): Participants were administered 0.07 mg CCH subcutaneously using a single injection technique. Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -22 and -1. Area 2 was administered CCH on Day -1.
  Interventions: Drug: Collagenase Clostridium Histolyticum Single Injection Technique
- Group 4: CCH Multiple Injection Technique (Experimental): Participants were administered 0.0653 mg CCH subcutaneously using a multiple injection technique.
  Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -43 and -22. Area 2 was administered CCH on Day -14.
  Interventions: Drug: Collagenase Clostridium Histolyticum Multiple Injection Technique
- Group 5: CCH Multiple Injection Technique (Experimental): Participants were administered 0.0653 mg CCH subcutaneously using a multiple injection technique.
  Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -24 and -3. Area 2 was administered CCH on Day -3.
  Interventions: Drug: Collagenase Clostridium Histolyticum Multiple Injection Technique
- Group 6: CCH Multiple Injection Technique (Experimental): Participants were administered 0.0653 mg CCH subcutaneously using a multiple injection technique.
  Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -22 and -1. Area 2 was administered CCH on Day -1.
  Interventions: Drug: Collagenase Clostridium Histolyticum Multiple Injection Technique

INTERVENTIONS:
Drug: Collagenase Clostridium Histolyticum Single Injection Technique — CCH was injected subcutaneously using a single injection technique. Dose per each administration was 0.07 mg.
  Other Names: EN3835; CCH
  Arms: Group 1: CCH Single Injection Technique; Group 2: CCH Single Injection Technique; Group 3: CCH Single Injection Technique
Drug: Collagenase Clostridium Histolyticum Multiple Injection Technique — CCH was injected subcutaneously using a multiple injection technique. Dose per each administration was 0.0653 mg.
  Other Names: EN3835; CCH
  Arms: Group 4: CCH Multiple Injection Technique; Group 5: CCH Multiple Injection Technique; Group 6: CCH Multiple Injection Technique

SUMMARY:
To evaluate the histopathology of subcutaneous tissue isolated after single or multiple Collagenase Clostridium Histolyticum (CCH) injection techniques in adult female participants undergoing abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Be adequately informed and understand the nature and risks of the study and be able to provide consent.
2. Be undergoing planned elective abdominoplasty.
3. Be willing to have their tissue donated for evaluation.
4. Be judged to be in good health.
5. Have a negative pregnancy test.
6. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the US Code of Federal Regulations (CFR) Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
2. Has systemic conditions (coagulation disorders, malignancy, keloidal scar, abnormal wound healing) that restricts study participation.
3. Has local (in the areas to be treated) conditions (thrombosis, vascular disorder, active infection/inflammation, active cutaneous alteration, tattoo/mole) that restricts study participation.
4. Required use of anticoagulant or antiplatelet medication (except ≤ 150 mg aspirin daily) before or during participation in the trial.
5. Past history of any abdominal surgery, including but not limited to: liposuction, caesarean section, appendectomy, cholecystectomy, or umbilical hernia repair.
6. Has used or intends to use any local applications/therapies/injections/procedures that restricts study participation.
7. Is presently nursing or providing breast milk in any manner.
8. Intends to become pregnant during the study.
9. Intends to initiate an intensive sport or exercise program regimen during the study.
10. Intends to use any tanning spray or tanning booths during the study.
11. Has received any investigational drug or treatment within 30 days prior to first injection of study drug.
12. Has a known systemic allergy to collagenase or any other excipient of study drug.
13. Has received any collagenase treatment at any time prior to treatment in this study.
14. Any other condition(s) that, in the investigator's opinion, might indicate the subject to be unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chajko, Study Director — Endo Pharmaceuticals
Locations (2):
- United States (2):
  - Endo Clinical Trial Site #1, Montclair, New Jersey
  - Endo Clinical Trial Site #2, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were divided among 6 different cohorts based on injection technique and respective dosing days. Two participants (Group 4 multiple injection technique) were not included in the Evaluable Population when their surgeries were delayed due to the effects of COVID-19 restrictions.
Groups:
- Group 1: Collagenase Clostridium Histolyticum (CCH) Single Injection Technique: Participants were administered 0.07 milligrams (mg) CCH subcutaneously using a single injection technique.
  Each participant had 2 marked areas of the abdomen (Area 1 and Area 2) selected for injection. Area 1 was administered CCH on Days -43 and -22. Area 2 was administered CCH on Day -14.
- Group 3: CCH Single Injection Technique: Participants were administered 0.07 mg CCH using a single injection technique. Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -22 and -1. Area 2 was administered CCH on Day -1.
Period: Overall Study
Arm/Group | Group 1: Collagenase Clostridium Histolyticum (CCH) Single Injection Technique | Group 2: CCH Single Injection Technique | Group 3: CCH Single Injection Technique | Group 4: CCH Multiple Injection Technique | Group 5: CCH Multiple Injection Technique | Group 6: CCH Multiple Injection Technique
Started | 2 | 1 | 1 | 4 | 1 | 1
Safety Population (All participants who received at least 1 injection of study drug irrespective of the timing window of abdominoplasty.) | 2 | 1 | 1 | 4 | 1 | 1
Evaluable Population (All participants who received at least 1 injection of study drug, underwent abdominoplasty within the protocol specified timelines, and had a histopathology and immunohistochemistry report.) | 2 | 1 | 1 | 2 | 1 | 1
Completed | 2 | 1 | 1 | 4 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least 1 injection of study drug irrespective of the timing window of abdominoplasty. Baseline characteristics (demographic) data were combined for all participants to protect personally identifiable information (PII) of the participant and to reduce risk of participant identification in the small population size of the 2 arms/groups.
Groups:
- CCH Subcutaneous Injection: Participants were administered 0.07 mg CCH using a single injection technique or 0.0653 mg CCH using a multiple injection technique.
Arm/Group | CCH Subcutaneous Injection
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Weight [Mean (Standard Deviation); unit: Kg] | 71.31 (16.275)
Height [Mean (Standard Deviation); unit: cm] | 164.47 (7.265)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.24 (4.460)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Histologic Change in a Tissue Specimen That Was Injected With CCH
Description: Tissue specimens isolated from participants undergoing an abdominoplasty procedure were observed for histopathological structure changes of tissues post treatment with CCH. The number of participants with a histologic change (as determined by the pathologist) in tissue dosed with CCH relative to control tissue (tissue not dosed with CCH) is reported.
Time Frame: Up to collection of the excised abdominal tissue on Day 0 (day of abdominoplasty)
Population: Evaluable Population: All participants who received at least 1 injection of study drug, underwent abdominoplasty within the protocol specified timelines, and had a histopathology and immunohistochemistry report.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: CCH Single Injection Technique: Participants were administered 0.07 mg CCH subcutaneously using a single injection technique.
  Each participant had 2 marked areas (Area 1 and Area 2) of the abdomen selected for injection. Area 1 was administered CCH on Days -43 and -22. Area 2 was administered CCH on Day -14.
Arm/Group | Group 1: CCH Single Injection Technique | Group 2: CCH Single Injection Technique | Group 3: CCH Single Injection Technique | Group 4: CCH Multiple Injection Technique | Group 5: CCH Multiple Injection Technique | Group 6: CCH Multiple Injection Technique
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 1 | 1
Participants | 2 | 1 | 1 | 2 | 1 | 1

2. Secondary Outcome: Number of Participants With a Histologic Change in a Tissue Specimen After 2 CCH Dose Injections Relative to a Tissue Specimen After 1 CCH Dose Injection
Description: Tissue specimens isolated from participants undergoing an abdominoplasty procedure were observed for histopathological structure changes of tissues post treatment with CCH. The number of participants with a histologic change (as determined by the pathologist) in a tissue specimen injected with 2 CCH dose injections (Treatment Area 1) relative to 1 CCH dose injection (Treatment Area 2) is reported.
Time Frame: Up to collection of the excised abdominal tissue on Day 0 (day of abdominoplasty)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: CCH Single Injection Technique | Group 2: CCH Single Injection Technique | Group 3: CCH Single Injection Technique | Group 4: CCH Multiple Injection Technique | Group 5: CCH Multiple Injection Technique | Group 6: CCH Multiple Injection Technique
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 1 | 1
Participants | 2 | 1 | 1 | 2 | 1 | 1

3. Secondary Outcome: Number of Participants With Anti-AUX-I and Anti-AUX-II Anti-Drug Antibodies (ADAs) After CCH Treatment
Description: Serum samples were analyzed for anti-AUX-I clostridial class I collagenase of ADAs and anti-AUX-II Clostridial class II collagenase of ADAs. The number of participants who developed anti-AUX-I and anti-AUX-II ADAs (positive ADA result) are reported.
Time Frame: End of Study (Day 28)
Population: Safety Population: All participants who received at least 1 injection of study drug irrespective of the timing window of abdominoplasty. ADA data is reported as overall population instead of individual groups due to the small number of participants per arm and to protect PII of the participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CCH Subcutaneous Injection
Number analyzed (Participants) | 10
Participants
  Anti-AUX-I ADAs | 9
  Anti-AUX-II ADAs | 5

4. Secondary Outcome: Number of Participants With Anti-AUX-I and Anti-AUX-II Neutralizing Antibodies (NAbs) After CCH Treatment
Description: Serum samples were analyzed for anti-AUX-I and Anti-AUX-II Nabs. The number of participants who developed anti-AUX-I and Anti-AUX-II NAbs (positive NAb results) are reported. Neutralizing antibodies were only tested from ADA positive participants.
Time Frame: End of Study (Day 28)
Population: All participants who received at least 1 injection of study drug and were positive for ADAs. NAb data is reported as overall analysis population instead of individual groups due to the small number of participants per arm and to protect PII of the participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CCH Subcutaneous Injection
Number analyzed (Participants) | 9
Participants
  Anti-AUX-I NAbs | 7
  Anti-AUX-II NAbs: number analyzed (Participants) | 5
  Anti-AUX-II NAbs | 3

ADVERSE EVENTS:
Time Frame: From first injection (earliest dosing visit at Day -43) up to collection of the excised abdominal tissue on Day 0 (day of abdominoplasty) for CCH injection treatment and up to end of study (Day 28 post-abdominoplasty surgery follow-up visit)
Description: Adverse events were collected throughout the study (up to Day 28 post-abdominoplasty surgery follow-up visit). Adverse events associated with local tolerability in treatment areas injected with CCH were collected up to the day abdominal tissue was excised.
Groups:
- Group 4: CCH Multiple Injection Technique: Participants were administered 0.0653 mg CCH subcutaneously using a multiple injection technique.
  Each participant had 2 marked (Area 1 and Area 2) areas of the abdomen selected for injection. Area 1 was administered CCH on Days -43 and -22. Area 2 was administered CCH on Day -14.
Arm/Group | Group 1: CCH Single Injection Technique | Group 2: CCH Single Injection Technique | Group 3: CCH Single Injection Technique | Group 4: CCH Multiple Injection Technique | Group 5: CCH Multiple Injection Technique | Group 6: CCH Multiple Injection Technique
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/4 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/4 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 4/4 | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: CCH Single Injection Technique (N=2) | Group 2: CCH Single Injection Technique (N=1) | Group 3: CCH Single Injection Technique (N=1) | Group 4: CCH Multiple Injection Technique (N=4) | Group 5: CCH Multiple Injection Technique (N=1) | Group 6: CCH Multiple Injection Technique (N=1)
Injection site oedema (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Injection site bruising (General disorders) | 1 | 1 | 1 | 3 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 4 | 1 | 1
Injection site haemorrhage (General disorders) | 2 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 4 | 1 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 4 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 3 | 1 | 1
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Post procedural erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 4 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This was considered an exploratory study by the Sponsor. No formal sample size calculations were performed. Completion of 8 participants provided minimal data to meet the primary objective in the evaluable population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04236635/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT04236635/SAP_001.pdf